CLINICAL TRIAL: NCT01164176
Title: An Open Label Multi-Center Phase II Study of RAD001 in Advanced Thyroid Cancer
Brief Title: Everolimus in Treating Patients With Locally Advanced or Metastatic Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2009-0542; YONSEI-CRAD001CKR12T; KCSG-HN-10-03
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-02

CONDITIONS: Head and Neck Cancer
Keywords: anaplastic thyroid cancer; insular thyroid cancer; recurrent thyroid cancer; stage III follicular thyroid cancer; stage III papillary thyroid cancer; stage IV follicular thyroid cancer; stage IV papillary thyroid cancer; thyroid gland medullary carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Thyroid Carcinoma, Anaplastic; Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary; Carcinoma, Medullary | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 group (Experimental)
  Interventions: Drug: everolimus; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: everolimus
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well everolimus works in treating patients with locally advanced or metastatic thyroid cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate response rate in patients with locally advanced or metastatic, unresectable or refractory thyroid cancer treated with everolimus.

Secondary

* To evaluate overall survival of these patients treated with everolimus.
* To evaluate progression-free survival of these patients.
* To evaluate toxicity of this therapy in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral everolimus once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for correlative studies.

After completion of study treatment, patients are followed up for 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed thyroid cancer

  * Progressive or refractory disease within the past 6 months
  * Locally advanced or metastatic disease
* Measurable disease, defined as ≥ 1 measurable lesion defined by RECIST criteria
* Not amenable to surgical resection or external-beam radiotherapy or refractory to radioiodine therapy
* No untreated brain metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Creatinine < 1.5 mg/dL
* Total bilirubin ≤ 1.0 times upper limit of normal (ULN)
* ALT and AST ≤ 3.0 times ULN
* No known hypersensitivity to the study drug
* No serious uncontrolled systemic intercurrent illness (e.g., infection or poorly controlled diabetes)
* No history of significant neurological or mental disorder, including seizures or dementia
* No other malignancy within the past 5 years except for carcinoma in situ of the cervix or nonmelanomatous carcinoma of the skin
* No active uncontrolled cardiac disease
* No myocardial infarction within the past 12 months
* Able to take oral medication
* No active peptic ulcer disease
* Must have patient compliance and geographic proximity for adequate follow-up

PRIOR CONCURRENT THERAPY:

* At least 30 days since prior mTor-inhibitor therapy (e.g., temsirolimus) or non-hormonal anticancer therapy
* At least 2 weeks since prior and no concurrent P-glycoprotein, CYP3A4, and CYP3A5 inhibitors or inducers
* No prior surgical procedure affecting absorption
* No other concurrent systemic chemotherapy, investigational drug, or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Response rate | every 3 month

SECONDARY OUTCOMES:
Overall survival | participants will be followed until death
Progression-free survival | participants will be followed until disease progression or death
Toxicity profile | participants will be followed until disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Byung Chul Cho, Principal Investigator — Yonsei University
Locations (7):
- South Korea (7):
  - Hallym University Sacred Heart Hospital, Anyang, Gyeonggi-do
  - Yeungnam University Medical Center, Daegu
  - National Cancer Center - Korea, Goyang
  - Kosin Medical Center Gospel Hospital, Pusan
  - Seoul National University Hospital, Seoul
  - Yonsei Cancer Center at Yonsei University Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul

REFERENCES:
- [Derived] Lim SM, Chang H, Yoon MJ, Hong YK, Kim H, Chung WY, Park CS, Nam KH, Kang SW, Kim MK, Kim SB, Lee SH, Kim HG, Na II, Kim YS, Choi MY, Kim JG, Park KU, Yun HJ, Kim JH, Cho BC. A multicenter, phase II trial of everolimus in locally advanced or metastatic thyroid cancer of all histologic subtypes. Ann Oncol. 2013 Dec;24(12):3089-94. doi: 10.1093/annonc/mdt379. Epub 2013 Sep 19. PMID 24050953